CLINICAL TRIAL: NCT04766489
Title: Evaluation of the Treatment Response in Breast Cancer Related Lymphedema After Mastectomy Surgery
Brief Title: Evaluation of the Treatment Response in Breast Cancer Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Göksel Tanıgör M.D., Researcher, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLUE-BCL
Record Dates: First submitted 2021-02-20; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Lymphedema of Upper Limb; Breast Cancer; Breast Cancer Lymphedema
Keywords: Lymphedema; Mastectomy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete Deongestive Therapy (Experimental): Patients will be given complete decongestive therapy for 5 days a week and for a mean of 20 sessions. Each session will be of approximately 2 hours and 15 minutes in duration, although short stretch bandaging will be left on for 23 hours a day.
  Interventions: Procedure: Complete Decongtestive Therapy

INTERVENTIONS:
Procedure: Complete Decongtestive Therapy — Patients will be given complete decongestive therapy, which includes decongestive exercises, manual lymphatic drainage, compression therapy(either through short stretch bandaging and/or pneumatic device) and exercise, for 5 days a week and for a mean of 20 sessions. Each session will be of 1 hour duration for compressive therapies(Short stretch bandages will be left on for 23 hours a day), 30 minutes of manual lymphatic drainage, and decongestive exercises 3 times a day for 15 minutes each time.
  Other Names: Aggresive treatment phase for lymphedema

SUMMARY:
This study aims to evaluate the effects of the treatment for breast cancer lymphedema. After taking a detailed history and giving a physical examination, breast cancer related lymphedema patients(n:30) will be informed and will be given Complete Decongestive Therapy, which includes decongestive exercises, manual lymphatic drainage, compression therapy(either through short stretch bandaging and/or pneumatic device) and exercise. Patients will be evaluated with limb volume, lymphedema index acquired through bioimpedance device, QuickDASH for upper extremity function, hand dynamometer for upper extremity grip strength and CLUE(Breast Cancer-Related Lymphedema of the Upper Extremity standardized clinical evaluation tool) scoring for lymphedema before and after the intervention. The values will be compared in order to show whether there are significant differences between before and after scores, and whether CLUE score is correlated with the other indicators of breast cancer related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lymphedema of the arm after mastectomy for breast cancer

Exclusion Criteria:

* Bilateral lymphedema
* Primary bone tumor and/or metastasis
* Patients with ongoing radiotherapy
* Circulation disorders of the upper extremity(eg; peripheral vascular disease, thrombosis)
* Patients with infectious lymphedema/elephantiasis
* Presence of local infection in upper extremities(cellulitis) and/or presence of severe systemic infection
* Carcinomatous lymphangitis
* Congestive heart failure(NYHA class 3 or 4)
* History of prosthesis on upper extremities
* Use of drugs which may alter the fluid or electrolyte balance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
CLUE score | 1 month
  Breast Cancer-Related Lymphedema of the Upper Extremity (CLUE) is a standardized clinical evaluation tool which was developed to evaluate the severity of the lymphedema, especially in the context of clinical trials. CLUE involves assessing obscuration of anatomical architecture (eg, bony prominences, tendons), deviation from normal anatomical contour, change of soft-tissue texture, and the presence of pitting or nonpitting edema. It consists of these four assessments conducted in three different parts or the upper extremity(arm, forearm and hand). CLUE scores have a range of 0 to 72, with greater numbers associated with more severe lymphedema. It was shown to be valid and reliable for the assessment of breast cancer related lymphedema by Spinelli et al.(1)

SECONDARY OUTCOMES:
Hand Grip Strength | 1 Month
  Hand grip strength: Hand grip strength will be measured using JAMAR® hand dynamometer. It has been used to assess hand grip strength in many studies over half a century. Patients will be asked to sit down with shoulder adducted, elbow flexed (90°) and forearm in the neutral position. Mean of the 3 measurements taken with 1 minute apart from each other will be recorded. Patients' measurements will be taken for both affected and unaffected arm, and will be recorded as kgf.
Extremity volume | 1 Month
  Volume measurements will be taken using ulnar styloid process as a index point, and circumferential measurements were taken with 5 cm spaces from distal to the proximal. Using a computer programme (Limb Volumes Professional version 5.0), the total volume of the arm will be calculated and recorded before and after the treatment for both arms.
  All patients' measurements will be taken by the same researcher, who happens to be experienced in this field.
Lymphedema index | 1 Month
  Lymphedema index will be acquired with a bioimpedance spectroscopy device (L-DEX U400, ImpediMed Limited, Brisbane-Australia). The device utilizes the characteristics of frequency dependent current flow to quantify changes in extracellular fluid in the patient's limb. The lymphedema index value increases on the scale with the higher levels of extracellular fluid, which is directly associated with the presence of lymphedema.
QuickDASH | 1 Month
  Short version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire(Quick-DASH) will be used to assess the function of the upper extremities. The Quick-DASH contains 11 items (scored 1-5) and reflects both function and pain in persons with musculoskeletal disorders of the upper extremity. To be able to calculate a score, at least 10 of the 11 items must be completed. The overall score ranges from 0 to 100 points with higher score representing greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plans of sharing data.

REFERENCES:
- [Result] Spinelli B, Kallan MJ, Zhang X, Cheville A, Troxel A, Cohn J, Dean L, Sturgeon K, Evangelista M, Zhang Z, Ebaugh D, Schmitz KH. Intra- and Interrater Reliability and Concurrent Validity of a New Tool for Assessment of Breast Cancer-Related Lymphedema of the Upper Extremity. Arch Phys Med Rehabil. 2019 Feb;100(2):315-326. doi: 10.1016/j.apmr.2018.08.185. Epub 2018 Oct 4. PMID 30291828